CLINICAL TRIAL: NCT06750640
Title: Acupoint Thermal Radiation Characteristics in Adolescents with Major Depressive Disorder and Establishment of Diagnostic Model
Brief Title: Acupoint Thermal Radiation Characteristics in Adolescents with MDD
Status: Completed | Type: Observational
Sponsor: Xiaomei Shao (Other)
Collaborators: Zhejiang Provincial Tongde Hospital (Other); First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor-Investigator, Xiaomei Shao, Prof, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Other Study IDs: 2022ZX010-IRT
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Major Depression
Keywords: Major Depression Disorder; acupoint temperature; adolescent
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Control group: There were 40 healthy control participants in the Healthy Control group.
  Interventions: Diagnostic Test: Infrared thermography
- Major Depression Disorder group: There were 60 MDD patients in the MDD group. All MDD adolescents received at least one IRT test. 26 MDD adolescents were detected by 2 investigators and 2 investigators both made 2 independent measurements in a week. 30 MDD subjects were detected the bilateral same name acupoint temperatures.
  Interventions: Diagnostic Test: Infrared thermography

INTERVENTIONS:
Diagnostic Test: Infrared thermography — A thermograph (NEC InfRec R450, Avio Infrared Technologies Co., Ltd., Tokyo) was used to record thermal images. The infrared camera was fixed on a tripod 1 m away from the subject to ensure that no shaking movements or vibrations occurred during the recording of thermal images. MDD related acupoints on the inner and outer sides of the limbs were detected. Appropriate body position was selected according to the different parts to be detected. Using the automatic interval saving shooting mode, one thermal picture was taken at 10-s intervals, 3 pictures were taken for each subject.

SUMMARY:
Modern studies have confirmed that skin temperature changes at acupoints when the body is under pathological conditions. This suggests that changes in the thermal radiation characteristics of acupoints can objectively respond to the symptoms of a disease. In this study, the investigators first evaluated reproducibility of acupoint temperature measurement by IRT. Secondly, the investigators explored the thermal radiation characteristics of MDD-related acupoints, built the diagnostic model for adolescent depression severity and the diagnostic model for MDD in adolescents based on acupoint temperature. Our research findings will provide new ideas, methods and visualisations for early screening, auxiliary diagnosis and condition assessment of MDD in adolescents.

DETAILED DESCRIPTION:
A total of 100 subjects were included, 60 adolescent with MDD (MDD group) and 40 healthy controls (HC group). All subjects accepted IRT detection.The random selection of 30 adolescent with MDD allowed the collection of the bilateral same name acupoint temperatures. Intra- and inter-observer reproducibility for the patients were examined in some randomly selected patients by 2 investigators and 2 investigators both made 2 independent measurements in a week. 30 MDD subjects were detected the bilateral same name acupoint temperatures.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the healthy control participants:

* 12years≤ age<18 years;
* SDS score <53;
* Adolescents with normal cognitive function can cooperate with the study;
* Adolescents and guardians agree to the study plan and sign the informed consent form.

Inclusion criteria for the major depression disorder participants:

* 12years≤ age<18 years;
* Self-rating Depression Scale (SDS) score ≥ 53;
* Language, cognition and communication ability are normal;
* Patients and guardians agree to the study plan and sign the informed consent form.

Exclusion Criteria:

Exclusion criteria both for the healthy control participants and major depression disorder participants:

* Severe anxiety, schizophrenia, or other serious mental illnesses;
* There are pigmentation, redness, infection or scarring on the skin at the site of detection;
* Patients with severe systemic diseases and their complications, serious infections, and major diseases of viscera, tissues, and systems;
* Female patients who were pregnant or lactating;
* Female patients who were during, or in proximity (±2 days) to their menstruation or ovulation;
* Patients with a body temperature ≥37.3°C;
* Inability to cooperate during the examination;
* Participating in any other clinical trials.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The diagnostic criteria of MDD were based on criteria proposed by the International Classification of Diseases 10th Edition (ICD-10). Healthy control participants were determined by a recent depression screening report for confirming their mental health conditions.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-03-05 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Acupoint emperature | Baseline
  Temperature of acupoints was measured by infrared thermography (IRT). IRT was not be performed on female subjects during their menstrual and ovulatory periods.

SECONDARY OUTCOMES:
The Self-Rating Depression Scale (SDS) Scores | Baseline
  The standard score is the total of all scores multiplied by 1.25 to the nearest whole number on this scale, which has 20 questions. A standard score below 53 is normal; 53-62 is mild depression; 63-72 is moderate depression; 72 or more is severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No